CLINICAL TRIAL: NCT01848041
Title: A Randomized, Double-Masked, Placebo-Controlled Phase 1/2a Study of the Efficacy and Safety of Two Dosing Regimens of RVL-1201 in the Treatment of Acquired Blepharoptosis
Brief Title: Safety and Efficacy Study of RVL-1201 in Acquired Blepharoptosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVL-1201-001
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Blepharoptosis
Keywords: Blepharoptosis; Ptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- RVL-1201 once daily (Experimental): RVL-1201 0.1% ophthalmic solution dosed one full drop per eye in the morning; one full drop of vehicle (placebo) per eye approximately 8 hours after the morning dose
  Interventions: Drug: RVL-1201
- RVL-1201 twice daily (Experimental): RVL-1201 0.1% ophthalmic solution dosed one full drop per eye BID; approximately 8 hours between the morning dose and the afternoon dose
  Interventions: Drug: RVL-1201
- RVL-1201 vehicle (placebo) (Placebo Comparator): RVL 1201 ophthalmic solution vehicle (placebo) dosed one full drop per eye BID; approximately 8 hours between the morning dose and the afternoon dose
  Interventions: Drug: RVL-1201 Vehicle Placebo

INTERVENTIONS:
Drug: RVL-1201 — RVL-1201 0.1% Ophthalmic Solution
  Other Names: Oxymetazoline Hydrochloride Ophthalmic Solution 0.1%
  Arms: RVL-1201 once daily; RVL-1201 twice daily
Drug: RVL-1201 Vehicle Placebo — RVL-1201 Vehicle Placebo
  Other Names: RVL-1201 Ophthalmic Solution 0.1% Placebo
  Arms: RVL-1201 vehicle (placebo)

SUMMARY:
This is an exploratory, proof of concept study to evaluate the safety and efficacy of RVL-1201 dosed once or twice daily for 14 days compared to a placebo (vehicle) control in patients with ptosis.

DETAILED DESCRIPTION:
This is an exploratory, proof-of-concept study. The objectives include establishing the efficacy and duration of effect of once daily (QD) or twice daily (BID) administration of RVL-1201 and the safety profile following 14 days of treatment in 72 subjects (24 per arm) with acquired blepharoptosis.

Efficacy will be assessed at each treatment visit by the Humphrey Visual Field 36-point ptosis protocol test, photographic measurement of marginal reflex distance, palpebral fissure distance and contrast sensitivity in the study eye only and Visual Acuity assessment in both eyes.

Safety assessments will include slit lamp examination/corneal fluorescein staining, pupil size measurement, ophthalmoscopy/ fundus examination, tonometry, visual acuity; urine pregnancy test (for women of childbearing potential only), vital signs (Heart Rate/Blood Pressure); and collection of adverse events. Subject rating of study medication comfort and assessment of ongoing tolerability will also be obtained.

Primary efficacy endpoint is the mean increase from baseline in points seen on the HVF 36-point ptosis protocol test at various timepoints according to a hierarchical analysis.

Analysis of exploratory endpoints will provide characterization of the efficacy and duration of effect of RVL-1201 with a variety of efficacy measures, as well as the potential additional effect of BID over QD dosing and safety profile of BID administration of RVL-1201. Exploratory endpoints will be analyzed by each regimen against placebo and between regimens and will include:

* The change from baseline in HVF, MRD, PFD, VA, and CS.
* The change from baseline in BP/HR

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects 18 years of age and older.
2. Presence of all of the following at Screening:

   1. Loss on HVF 36-point ptosis protocol test of ≥ 8 points in points not seen at or above 10° from fixation in the superior visual field; AND
   2. Marginal reflex distance (MRD), the distance from the central pupillary light reflex to the upper lid margin, of ≤ 2.5 mm in the same eye as Inclusion Criterion #2a; AND
   3. Corrected Snellen visual acuity (VA) of 20/40 or better (refraction must be within 6 months of Visit 1) in the same eye as Inclusion Criteria #2a and #2b.
3. No contraindications for treatment of both eyes as specified in Exclusion Criteria #1-14.
4. Female subjects must be 1-year postmenopausal, surgically sterilized, or women of childbearing potential with a negative urine pregnancy test at Visit 1. Women of childbearing potential must use an acceptable form of contraception throughout the study.
5. Provide informed consent prior to undergoing any study-related procedures.

Exclusion Criteria:

In either eye:

1. Congenital ptosis
2. Pseudoptosis
3. Horner syndrome
4. Marcus Gunn jaw-winking syndrome
5. Myasthenia gravis
6. Mechanical ptosis, including ptosis due to orbital or lid tumor, cicatricial processes affecting the movements of the upper lid, and enophthalmos
7. Dermatochalasis as the sole cause of the signs of ptosis
8. Previous ptosis surgery
9. Lid position affected by lid or conjunctival scarring
10. Current use of prescribed dry eye medication or punctal plugs; artificial tears are allowed
11. Visual field loss from any cause other than ptosis
12. Inability to fixate on the central fixation target of the HVF
13. Primary open-angle glaucoma or ocular hypertension, intraocular pressure (IOP) > 24 mm Hg, or current use/use within 1 month prior to Visit 1 of any antiglaucoma medications.
14. History of closed/narrow angle glaucoma (unless patent peripheral iridotomy has been performed > 3 months prior to Visit 1 and IOP < 20 mm Hg) or normal-tension glaucoma
15. Use of over-the-counter vasoconstrictor/decongestant eye medication (eg, Visine® L.R.®) or any α-adrenergic agonist (including OTC products) at any time during the study
16. Contact lens wear during the study period

    General:
17. Resting heart rate (HR) outside the normal range (60 - 100 beats per minute)
18. Hypertension diastolic blood pressure (BP) > 105 mm Hg
19. Use of monoamine oxidase inhibitors (MAOIs; eg, isocarboxazid, phenelzine, tranylcypromine) within 14 days prior to Visit 1 or during the study
20. Use of beta blockers (eg, propranolol, metoprolol, labetalol) within 14 days prior to Visit 1 or during the study
21. Use of maprotiline, selective serotonin reuptake inhibitors ([SSRIs] eg, citalopram, escitalopram, paroxetine, fluoxetine, fluvoxamine, sertraline) or tricyclic antidepressants (eg, amitriptyline, doxepin, nortriptyline, amoxapine, clomipramine, desipramine, imipramine, protriptyline, trimipramine) at any time during the study
22. A history of myocardial infarction, angina, arrhythmia, or irregular pulse
23. Advanced arteriosclerotic disease
24. History of thyroid disease
25. Insulin-dependent diabetes or diabetes requiring oral hypoglycemic drugs; diet-controlled diabetes is allowed
26. Pregnancy or lactation
27. Diagnosed benign prostatic hypertrophy requiring medicinal therapy.
28. History of contact or systemic allergic reaction to oxymetazoline or other sympathomimetic drugs (eg, phenylephrine, pseudoephedrine, ephedrine, phenylpropanolamine, fepradinol, or methoxamine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chuck Slonim, MD, Principal Investigator — Oculos Clinical Research
Locations (1):
- Morrow, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RVL-1201 QD: RVL-1201 0.1% ophthalmic solution dosed one full drop per eye in the morning; one full drop of vehicle (placebo) per eye approximately 8 hours after the morning dose
  RVL-1201: RVL-1201 0.1% Ophthalmic Solution
- RVL-1201 BID: RVL-1201 0.1% ophthalmic solution dosed one full drop per eye BID; approximately 8 hours between the morning dose and the afternoon dose
  RVL-1201: RVL-1201 0.1% Ophthalmic Solution
- RVL-1201 Vehicle (Placebo) BID: RVL 1201 ophthalmic solution vehicle (placebo) dosed one full drop per eye BID; approximately 8 hours between the morning dose and the afternoon dose
  RVL-1201 Vehicle Placebo: RVL-1201 Vehicle Placebo
Period: Overall Study
Arm/Group | RVL-1201 QD | RVL-1201 BID | RVL-1201 Vehicle (Placebo) BID
Started | 15 | 16 | 15
Completed | 15 | 16 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | RVL-1201 QD | RVL-1201 BID | RVL-1201 Vehicle (Placebo) BID | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 13 | 10 | 31
  >=65 years | 7 | 3 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.33) | 58.7 (10.47) | 58.3 (11.23) | 60.4 (10.80)
Age, Customized [Median (Full Range); unit: years] | 63 [40 to 78] | 60 [34 to 75] | 60 [33 to 73] | 61.5 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 11 | 34
  Male | 2 | 6 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 9 | 29
  Not Hispanic or Latino | 4 | 7 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 15 | 14 | 12 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 15 | 46
Iris Color OD/OS [Count of Participants; unit: Participants] — Right Eye (OD), Left Eye (OS)
  Participants
    Iris Color OD: Blue | 4 | 4 | 1 | 9
    Iris Color OD: Brown | 10 | 11 | 13 | 34
    Iris Color OD: Green | 0 | 1 | 1 | 2
    Iris Color OD: Hazel | 1 | 0 | 0 | 1
    Iris Color OD: Grey | 0 | 0 | 0 | 0
    Iris Color OD: Other | 0 | 0 | 0 | 0
    Iris Color OS: Blue | 4 | 4 | 1 | 9
    Iris Color OS: Brown | 10 | 11 | 13 | 34
    Iris Color OS: Green | 0 | 1 | 1 | 2
    Iris Color OS: Hazel | 1 | 0 | 0 | 1
    Iris Color OS: Grey | 0 | 0 | 0 | 0
    Iris Color OS: Other | 0 | 0 | 0 | 0
Lens Status OD/OS [Count of Participants; unit: Participants] — Lens Status of Phakic (implanted together with the natural), Aphakic (missing) or Pseudophakic (false - meaning not natural) is the type of eye lens. Right Eye (OD), Left Eye (OS)
  Participants
    Lens Status OD: Phakic, a person with an intact natural lens | 9 | 11 | 11 | 31
    Lens Status OD: Aphakic, a person with a natural lens was extracted and no intraocular lens was implanted. | 0 | 0 | 0 | 0
    Lens Status OD: Pseudophakic, a person who has had a lens extracted and an intraocular lens placed | 6 | 5 | 4 | 15
    Lens Status OS: Phakic, a person with an intact natural lens | 9 | 12 | 11 | 32
    Lens Status OS: Aphakic, a person with a natural lens was extracted and no intraocular lens was implanted. | 0 | 0 | 0 | 0
    Lens Status OS: Pseudophakic, a person who has had a lens extracted and an intraocular lens placed | 6 | 4 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Humphrey Visual Field
Description: The mean change from baseline (Day 0, Hour 0) in number of points seen on the HVF 36-point ptosis protocol test according to a pre-planned hierarchical analysis as follows:
  1. Hour 6 on Visit 4 (Day 13) for the BID regimen versus vehicle
  2. Hour 6 on Visit 4 (Day 13) for the QD regimen versus vehicle
  3. Hour 2 on Visit 4 (Day 13) for the BID regimen versus vehicle
  4. Hour 2 on Visit 4 (Day 13) for the QD regimen versus vehicle
  Testing was performed using a Humphrey perimeter at a grid of 36 points confined to the superior hemifield extending 55° to either side of fixation and 45° superior to fixation. Testing was accomplished in the standard fashion using a varying 4-mm2 or 5-mm2 stimulus to determine the visual sensitivity for each grid point in the field (Riemann et al, 2000). A 4-mm2 stimulus was acceptable, but a 5-mm2 stimulus was preferred, if available.
Time Frame: Baseline (Day 0, Hour 0), Visit 4 (Day 13, Hour 2) and Visit 4 (Day 13, Hour 6)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Points seen
Arm/Group | RVL-1201 Once Daily | RVL-1201 Twice Daily | RVL-1201 Vehicle (Placebo)
Number analyzed (Participants) | 15 | 16 | 15
Points seen
  Base Line (Day 0, Hour 0): number analyzed (Participants) | 15 | 14 | 15
  Base Line (Day 0, Hour 0) | 9.8 (5.07) | 12.1 (4.64) | 11.1 (4.74)
  Visit 4 (Day 13, Hour 2): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 2) | 16.1 (5.35) | 15.7 (4.63) | 15.7 (5.64)
  Visit 4 (Day 13, Hour 6) | 15.9 (5.29) | 17.0 (4.51) | 17.1 (5.02)

2. Secondary Outcome: Marginal Reflex Distance
Description: Change from baseline in MRD by regimen against placebo and between regimen.
  The distance from the pupillary light reflex to the central margin of the upper eyelid is the MRD. The MRD will be measured from the external photograph using calipers and the millimeter ruler as the legend.
Time Frame: Baseline (Day 0, Hour 0), Visit 4 (Day 13, Hour 2) and Visit 4 (Day 13, Hour 6)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | RVL-1201 Once Daily | RVL-1201 Twice Daily | RVL-1201 Vehicle (Placebo)
Number analyzed (Participants) | 15 | 16 | 15
Millimeters (mm)
  Baseline (Day 0, Hour 0): number analyzed (Participants) | 15 | 14 | 15
  Baseline (Day 0, Hour 0) | 1.6 (0.77) | 1.6 (0.84) | 1.6 (0.63)
  Visit 4 (Day 13, Hour 2): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 2) | 2.4 (0.99) | 2.3 (1.19) | 2.0 (0.95)
  Visit 4 (Day 13, Hour 6): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 6) | 2.4 (1.00) | 2.5 (1.13) | 2.2 (1.07)

3. Secondary Outcome: Palpebral Fissure Distance Measurement
Description: Change from baseline in PFD by regimen against placebo and between regimen.
  The PFD is the distance from the upper lid margin to the lower lid margin measured through the central visual axis. It will be measured from the external photograph using handheld calipers and the millimeter ruler as the legend.
Time Frame: Baseline (Day 0, Hour 0), Visit 4 (Day 13, Hour 2) and Visit 4 (Day 13, Hour 6)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | RVL-1201 Once Daily | RVL-1201 Twice Daily | RVL-1201 Vehicle (Placebo)
Number analyzed (Participants) | 15 | 16 | 15
Millimeters (mm)
  Baseline (Day 0, Hour 0): number analyzed (Participants) | 15 | 14 | 15
  Baseline (Day 0, Hour 0) | 6.2 (1.16) | 6.5 (1.10) | 6.5 (1.55)
  Visit 4 (Day 13, Hour 2): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 2) | 6.9 (1.35) | 7.1 (1.72) | 6.6 (1.67)
  Visit 4 (Day 13, Hour 6): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 6) | 7.0 (1.51) | 7.5 (1.45) | 6.8 (1.35)

4. Secondary Outcome: Contrast Sensitivity
Description: Change from baseline in CS by regimen against placebo and between regimen.
  The Pelli-Robson contrast sensitivity chart will be used at a distance of 1 meter. The subject was instructed to begin reading the letters at the top of the chart and to continue reading across and down the chart. Testing was discontinued when 2 of 3 letters were named incorrectly. The test was scored using the letter-by-letter method where a value of 0.05 log CS is given per correct letter (Haymes et al, 2006).
Time Frame: Baseline (Day 0, Hour 0), Visit 4 (Day 13, Hour 2) and Visit 4 (Day 13, Hour 6)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Letters Read
Arm/Group | RVL-1201 Once Daily | RVL-1201 Twice Daily | RVL-1201 Vehicle (Placebo)
Number analyzed (Participants) | 15 | 16 | 15
Letters Read
  Baseline (Day 0, Hour 0): number analyzed (Participants) | 15 | 14 | 15
  Baseline (Day 0, Hour 0) | 33.1 (4.05) | 34.7 (6.14) | 33.3 (5.81)
  Visit 4 (Day 13, Hour 2): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 2) | 34.7 (4.45) | 35.8 (4.28) | 35.3 (4.79)
  Visit 4 (Day 13, Hour 6): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 6) | 35.5 (3.81) | 36.8 (3.29) | 35.1 (4.18)

5. Secondary Outcome: Corrected Snellen Visual Acuity
Description: Change from baseline in VA by regimen against placebo and between regimen.
  Corrected Snellen VA measurement was performed with the Snellen eye chart using subjects current corrective lens prescription at a distance equivalent to 20 feet (6 meters).
Time Frame: Baseline (Day 0, Hour 0), Visit 4 (Day 13, Hour 2) and Visit 4 (Day 13, Hour 6)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | RVL-1201 QD | RVL-1201 BID | RVL-1201 Vehicle (Placebo) BID
Number analyzed (Participants) | 15 | 16 | 15
LogMAR
  Baseline (Day 0, Hour 0): number analyzed (Participants) | 15 | 14 | 15
  Baseline (Day 0, Hour 0) | 0.071 (0.0859) | 0.086 (0.0988) | 0.081 (0.0770)
  Visit 4 (Day 13, Hour 2): number analyzed (Participants) | 15 | 14 | 15
  Visit 4 (Day 13, Hour 2) | 0.055 (0.0739) | 0.024 (0.1043) | 0.059 (0.1190)
  Visit 4 (Day 13, Hour 6) | 0.026 (0.0891) | 0.023 (0.0949) | 0.053 (0.1018)

ADVERSE EVENTS:
Time Frame: 14 Days
Description: AEs were those with onset after randomization or if occurring prior to randomization, that worsened after randomization.
Arm/Group | RVL-1201 QD | RVL-1201 BID | RVL-1201 Vehicle (Placebo) BID
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 5/16 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 QD (N=15) | RVL-1201 BID (N=16) | RVL-1201 Vehicle (Placebo) BID (N=15)
Punctate keratitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Ocular Discomfort (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Instillation Site Dryness (General disorders) | 1 (2) | 0 (0) | 0 (0)
Instillation Site Foreign Body Sensation (General disorders) | 1 (2) | 2 (4) | 0 (0)
Instillation Site Pruritus (General disorders) | 1 (4) | 1 (2) | 0 (0)
Instillation Site Pain (General disorders) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes